CLINICAL TRIAL: NCT06836492
Title: A Prospective Clinical Cohort Study on Stratified Treatment of Rhabdomyosarcoma Based on Risk Factors: a Single Arm Trial.
Brief Title: A Prospective Clinical Cohort Study on Stratified Treatment of Rhabdomyosarcoma Based on Risk Factors.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yizhuo Zhang (Other)
Responsible Party: Sponsor-Investigator, Yizhuo Zhang, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-RMS
Record Dates: First submitted 2023-08-08; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Rhabdomyosarcoma; Pediatric Cancer
MeSH Terms: conditions — Rhabdomyosarcoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low risk (Other)
  Interventions: Combination Product: VAC，VAC/VII，CAV/IE
- Moderate risk (Other)
  Interventions: Combination Product: VAC，VAC/VII，CAV/IE
- High risk (Other)
  Interventions: Combination Product: VAC，VAC/VII，CAV/IE
- Very high risk (Other)
  Interventions: Combination Product: VAC，VAC/VII，CAV/IE

INTERVENTIONS:
Combination Product: VAC，VAC/VII，CAV/IE — Low risk: VAC Intermediate risk: VAC/VII High risk: CAV/IE Very high risk: CAV/VIP

SUMMARY:
The purpose is to explore the efficacy and safety of the SYSUCC-RMS regimen for pediatric RMS patients and to explore the impact of concurrent radiotherapy and chemotherapy on the survival rate of low-risk, medium risk, high-risk, and extremely high-risk patients in children.

ELIGIBILITY:
Inclusion Criteria:

1. 0 years < age < 18 years old, regardless of gender;
2. Tumor patients diagnosed by histopathology or bone marrow cytology;
3. Patients are treated for the first time;
4. ECoG score ≤ 2;
5. The expected survival time is more than 8 months;
6. Patient's parent or guardian signs informed consent.

Exclusion Criteria:

1. Combined with immunodeficiency disease
2. Second tumor

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The objective response rate (ORR) | Up to 1 year
  The ORR was calculated based on the best overall response.
disease control rate (DCR) | Up to 1 year
progression-free survival (PFS) | Up to 10 years
  Furthermore, we provided Kaplan-Meier plots for PFS
overall survival (OS) | Up to 10 years
  Furthermore, we provided Kaplan-Meier plots for OS.

SECONDARY OUTCOMES:
The safety of the SYSUCC-RMS regimen for pediatric RMS patients. | Up to 10 years
  Toxicity will be evaluated according to the Common Terminology Criteria for Adverse Event (CTC AE) scale, version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Suying Lu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No